CLINICAL TRIAL: NCT03640013
Title: A Randomized Clinical Trial Comparing Hall vs Conventional Technique in Placing Preformed Metal Crowns From Sudan
Brief Title: Comparing Hall vs Conventional Technique in Placing Preformed Metal Crowns From Sudan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khartoum Centre for Research and Medical Training (Other)
Responsible Party: Principal Investigator, Fadil Elamin, Principal Investigator, Khartoum Centre for Research and Medical Training
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KhartoumCentre
Record Dates: First submitted 2018-08-12; First posted 2018-08-21 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Controlled randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Technique (Experimental): The intervention involves removal from the primary molar and a preformed metal crown is placed using glass ionomer. The subject is then asked to bite until crown is seated. No occlusal adjustment is carried out.
  Interventions: Procedure: Hall Technique PMC
- Conventional Technique (Other): The procedure involves administering local anesthetic and the intervention involves remoal of caries from the affected primary molar. The tooth is then reshaped and contoured to to enable a preformed metal crown placement. Occlusal and marginal fit is improved by crimping the metal crown to improve fit. The preformed metal crown is cemented with glass ionomer restorative material and occlusion finally checked. The subject is then asked to bite on a cotton roll for two minutes until the cement has set.
  Interventions: Procedure: Hall Technique PMC

INTERVENTIONS:
Procedure: Hall Technique PMC — Hall Technique primary fitted crowns to restore carious primary molars

SUMMARY:
Preformed metal crowns (PMCs) have high success rates in restoring primary molars in children but they were not generally used by dentists, especially in developing countries due to its demand of high clinical skills with the conventional technique (CT). The biological approach, Hall technique (HT), requires less training and can be placed by less experienced dental operators including therapists. Previous studies were mainly carried out in developed countries. The aims were to investigate and compare the efficacies and cost-effectiveness of PMCs placed by these two techniques.

DETAILED DESCRIPTION:
A prospective randomised control trial design was used. The study was carried out in a dental practice in Sudan, an under-developed country with lower social economic group. Children between 5-8 years were invited and selected if they met the inclusion criteria. Only those who had 1-2 carious primary molars needing PMCs were randomised. The PMCs were placed by a dentist in the CT arm and by a therapist in the HT arm. The children were follow up every 6 months up to 2 years. The demographic details, periodontal health, occlusion, children anxieties, and procedure time were recorded. The Kaplan-Meier survival rates for each arm were calculated. The incremental cost effectiveness ratio (ICER) was calculated using the results and the local salaries

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with Class I or class II carious primary molars

Exclusion Criteria:

* Had a compromised medical history
* Were pre- or un-cooperative to have clinical examinations
* Lived in remote villages and were unlikely to return for follow-up
* Had teeth with pain or sepsis
* Had teeth with caries extended in pulp either from clinical or radiographic examinations

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Survival | 24 months
  If PMC intact and crown functional or not

SECONDARY OUTCOMES:
Gingival helath | 24 months
  Modified gingival index after Löe et al. (1967); Scale; 0=No disease; 1=hyperplasia with no bleeding; 2= hyperplasia with bleeding
Plaque Index | 24 months
  Plaque accumulation around preformed metal crown after Loe et al (1967); Scale: 0= no plaque, 1= subgingival plaque; 2= supragingival plaque
Occlusion | 24 months
  Natural teeth are in occlusion following PMC placement
Anxiety | 12 months
  Self perceived anxiety using facial image scale after Buchanan and Niven (2002) using 5 facial diagrams ranging from sad to smiley faces: Scale; 1-5; 1=extremely happy to 5=extremely unhappy

CONTACTS AND LOCATIONS:
Overall Officials: Dr Yousra, PhD, Study Director — University of Khartoum

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Innes NP, Ricketts D, Chong LY, Keightley AJ, Lamont T, Santamaria RM. Preformed crowns for decayed primary molar teeth. Cochrane Database Syst Rev. 2015 Dec 31;2015(12):CD005512. doi: 10.1002/14651858.CD005512.pub3. PMID 26718872
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Buchanan H, Niven N. Validation of a Facial Image Scale to assess child dental anxiety. Int J Paediatr Dent. 2002 Jan;12(1):47-52. PMID 11853248
- [Derived] Elamin F, Abdelazeem N, Salah I, Mirghani Y, Wong F. A randomized clinical trial comparing Hall vs conventional technique in placing preformed metal crowns from Sudan. PLoS One. 2019 Jun 3;14(6):e0217740. doi: 10.1371/journal.pone.0217740. eCollection 2019. PMID 31158253